CLINICAL TRIAL: NCT00326989
Title: Extracorporal Shock Wave Therapy for Induction of Therapeutic Neovascularization and Homing of Bone Marrow Progenitor Cells in Patients With Chronic Ischemic Heart Disease
Brief Title: Cell-Wave Study: Combined Extracorporal Shock Wave Therapy and Intracoronary Cell Therapy in Chronic Ischemic Myocardium
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, A. M. Zeiher, Prof. Dr. Andreas M. Zeiher, Johann Wolfgang Goethe University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2005-005709-50; Cellwave CHF
Record Dates: First submitted 2006-05-16; First posted 2006-05-17 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Congestive Heart Failure
Keywords: Extracorporal shock wave therapy; Cell therapy
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Low-dose shock wave treatment & Placebo (Active Comparator)
  Interventions: Procedure: intracoronary stem cell therapy
- low-dose shock-wave treatment & Cell therapy (Active Comparator)
  Interventions: Procedure: intracoronary stem cell therapy
- High-dose shock-wave treatment & Placebo (Active Comparator)
  Interventions: Procedure: intracoronary stem cell therapy
- High-dose shock-wave treatment & cell therapy (Active Comparator)
  Interventions: Procedure: intracoronary stem cell therapy
- Placebo shock-wave treatment & cell therapy (Active Comparator)
  Interventions: Procedure: intracoronary stem cell therapy

INTERVENTIONS:
Procedure: intracoronary stem cell therapy — extracorporal shock waves prior to intracoronary cell therapy

SUMMARY:
Extracorporal shock wave therapy is performed prior to cell therapy for induction of therapeutic neovascularization and improvement of homing of bone marrow progenitor cells in patients with chronic ischemic heart disease following anterior myocardial infarction.

Shock waves can induce growth factor expression in the ischemic myocardium and might augment homing of autologous bone marrow mononuclear cells which are injected intracoronary 24 h following shock wave therapy

DETAILED DESCRIPTION:
Single center, Phase I-II Study (Safety, Feasibility and Efficacy) Double-blind, randomised trial (Cell therapy), single blind (Shockwave)

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic ischemic heart disease
* Patients with anterior myocardial infarction > 3months
* EF < 50% or NYHA II-IV
* Age 18-80
* Informed consent

Exclusion Criteria:

* Ventricular thrombus
* Infarct < 3 months.
* Active infection or fever
* Chronic inflammatory disease (e.g M. Crohn, Rheumatoid Arthritis)
* HIV Infection oder active Hepatitis
* Neoplastic disease w/o complete remission within 5 years
* Stroke < 3months
* Creatinine > 2 mg/dl
* Relevant Liver disease (GOT > twice the upper limit).
* Anemia (Hemoglobin <10 mg/dl)
* Thrombocytopenia < 100.000/µl
* Allergies to Aspirin, Clopidogrel, Heparin
* History of bleeding disorder
* History of coagulopathy
* Gastrointestinal Bleeding < 3 months
* Surgery or Trauma < 2 months
* Pregnancy
* Mental Retardation
* Participation in other clinical study < 1 month

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2006-05; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Improvement in global ejection fraction on LV angiography | 4 months

SECONDARY OUTCOMES:
Global or regional wall motion at 4 months and 1 year | 4 months
NYHA Class | 4 months
NT BNP levels | 4 months
MACE | 4 months
Life quality | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Andreas M Zeiher, MD, Principal Investigator — Div. of Cardiology, University of Frankfurt, Germany; Dirk H Walter, MD, Study Director — Div. of Cardiology, University of Frankfurt
Locations (1):
- Div. of Cardiology , University of Frankfurt, Frankfurt, Germany

REFERENCES:
- [Derived] Assmus B, Walter DH, Seeger FH, Leistner DM, Steiner J, Ziegler I, Lutz A, Khaled W, Klotsche J, Tonn T, Dimmeler S, Zeiher AM. Effect of shock wave-facilitated intracoronary cell therapy on LVEF in patients with chronic heart failure: the CELLWAVE randomized clinical trial. JAMA. 2013 Apr 17;309(15):1622-31. doi: 10.1001/jama.2013.3527. PMID 23592107
- [Derived] Leistner DM, Seeger FH, Fischer A, Roxe T, Klotsche J, Iekushi K, Seeger T, Assmus B, Honold J, Karakas M, Badenhoop K, Frantz S, Dimmeler S, Zeiher AM. Elevated levels of the mediator of catabolic bone remodeling RANKL in the bone marrow environment link chronic heart failure with osteoporosis. Circ Heart Fail. 2012 Nov;5(6):769-77. doi: 10.1161/CIRCHEARTFAILURE.111.966093. Epub 2012 Aug 30. PMID 22936827